CLINICAL TRIAL: NCT05714982
Title: Randomized Clinical Trial Evaluating the Impact of E-cigarette Device Warnings
Brief Title: Impact of E-cigarette Device Warnings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 21-0469; R01DA048390 (NIH)
Record Dates: First submitted 2023-01-24; First posted 2023-02-06 (Actual); Results first posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-08

CONDITIONS: Vaping Behaviors
Keywords: Vaping; Tobacco use; E-cigarette use
MeSH Terms: conditions — Vaping; Tobacco Use | interventions — Drug Labeling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Label with text health warning (Experimental): Labels with e-cigarette health warning that include text about health harms of vaping will be applied to participants' vaping devices and refills.
  Interventions: Other: Label with text health warning
- Label with pictorial health warning (Experimental): Labels with e-cigarette health warning that include the same text about health harms of vaping and corresponding pictorial images will be applied to participants' vaping devices and refills.
  Interventions: Other: Label with pictorial health warning
- Label with neutral statements about vaping (Other): Labels with neutral statements about vaping will be applied to participants' vaping devices and refills.
  Interventions: Other: Label with neutral statements about vaping

INTERVENTIONS:
Other: Label with text health warning — Labels with e-cigarette health warning that include text about health harms of vaping will be applied to participants' vaping devices and refills. At Visit 1, devices and refills will be labeled with 2 warnings based on their assigned trial arm; at Visit 3, they will get 2 additional warnings based on their assigned trial arm. The order of the 4 labels within this trial arm will be randomized using a Latin square design. Study investigators developed the text and design of these labels.
  Arms: Label with text health warning
Other: Label with pictorial health warning — Labels with e-cigarette health warning that include the same text about health harms of vaping and corresponding pictorial images will be applied to participants' vaping devices and refills. At Visit 1, devices and refills will be labeled with 2 warnings based on their assigned trial arm; at Visit 3, they will get 2 additional warnings based on their assigned trial arm. The order of the 4 labels within this trial arm will be randomized using a Latin square design. Study investigators developed the text and design of these labels.
  Arms: Label with pictorial health warning
Other: Label with neutral statements about vaping — Labels with neutral statements about vaping will be applied to participants' vaping devices and refills. At Visit 1, devices and refills will be labeled with 2 statements based on their assigned trial arm; at Visit 3, they will get 2 additional statements based on their assigned trial arm. The order of the 4 labels within this trial arm will be randomized using a Latin square design. Study investigators developed the text and design of these labels.
  Arms: Label with neutral statements about vaping

SUMMARY:
The purpose of this randomized clinical trial is to determine whether e-cigarette warnings increase intentions to quit vaping without the unintended consequence of pushing users toward smoking. This trial addresses these issues by evaluating the impact of e-cigarette warnings by randomly assigning vapers to have their devices and refills labeled with control messages, text warnings, or pictorial warnings. Participants will be US adult (ages 21+) vapers. The trial expects ~1,200 participants to complete Visits 1, 3, and 5.

DETAILED DESCRIPTION:
This trial will assess the impact of e-cigarette warnings on vapers' devices and refills in a randomized clinical trial.

Recruitment: Vapers will first undergo screening online or call the study center to complete the screening survey over the phone. Trial staff will schedule eligible vapers for 2 in-person visits. For each of the 2 visits, vapers will be asked to bring the vapes and refill materials they plan to use over the next 2 weeks.

Informed Consent: Prior to consenting vapers, trial staff will visually inspect photo identification of vapers to confirm that they are 21 years or older. At the beginning of the first appointment, trial staff will explain the consent form and ask the vaper to read the form. Once the participant has finished reading the form, the trial staff member will ask the participant if he or she has any questions. Then both parties will sign the consent form and the participant will receive a copy of the consent form.

Randomization: At the first visit, trial staff will randomly assign participants to one of the three trial arms by using Qualtrics software. Vapers have an equal chance of being randomized to have labels with control, text, or pictorial warnings.

Assessment: Participants will attend 2 in-person appointments at the study office (at Visit 1 and Visit 3 that are spaced 2 weeks apart). The visits will last about 45-60 minutes. At Visit 1 participants will take a survey, have their vape device and refills labeled based on their trial arm, and take another survey. At Visit 3, participants take a survey and have their vape device and refills labeled based on their trial arm. Participants will also be e-mailed 3 more surveys to complete online at home (taken at Visit 2, 4, and 5). Thus participants will take 5 weekly surveys overall.

Detailed description of the intervention: At each in-person appointment, participants will bring in the vapes and refills they plan to use over the next 2 weeks for labeling. While participants are taking the survey, trial staff will label the devices and refills based on their trial arm.

Participants randomized to the text warning arm will have labels with information about the health harms of vaping applied to their vapes and refills. Participants randomized to the pictorial arm will have labels with pictorial images and text about the health harms of vaping. Participants assigned to the control arm will have labels with neutral statements about vaping. Each trial arm will have four labels (two labels for Visit 1 and two additional labels for Visit 3). Trial staff will return labeled vapes and refills in a clear plastic bag with the e-cigarette warning labels applied to a card. Trial investigators developed the text, images, and design of these labels.

The trial staff will instruct participants in all trial arms to vape or not vape as they normally would. At the end of the trial, participants will receive a link to more information about the risks of vaping and tobacco use.

ELIGIBILITY:
Inclusion Criteria:

* Be 21 years or older
* Currently vape every day or some days
* Use an e-cigarette that contains nicotine
* Be able to attend 2 in-person appointments
* Be able to bring in e-cigarette device and 2 weeks' worth or refills to 2 in-person appointments
* Be willing to let us apply a sticker to the device and refill materials
* Be willing to use only the labeled e-cigarette during the study
* Be able to complete 3 surveys online at home
* Be able to read and speak English
* Be able to complete a survey on a computer without help

Exclusion Criteria:

* Pregnant people
* If e-cigarette device cannot be labeled
* Vapers concurrently enrolled in any research studies about vaping or using other tobacco products
* Vapers who live in the same household as someone who has enrolled in the study

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1369 (Actual)
Dates: Start 2023-02-23 (Actual); Primary Completion 2024-07-23 (Actual); Study Completion 2024-07-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Noel Brewer, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Ewald & Wasserman Research Consultants, LLC, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The trial investigators will produce a de-identified dataset and codebook for sharing with external investigators, making use of the UNC Dataverse digital data repository (dataverse.unc.edu) hosted by the Odum Institute Data Archive.
Supporting Information: SAP, Analytic Code
Time Frame: The data will be available beginning 12 to 36 months following the primary publication.
Access Criteria: To obtain a copy of the dataset and codebook, a research scientist will have to submit a request in writing, identifying themselves and their affiliated institution, indicating what they plan to do with the data, and including assurances that they will not share the data with others without the written permission of the PI. Requestors must already have institutional review board, independent ethics committee, or research ethics board approval as applicable. Requestors must obtain a data use agreement through UNC's Office of Industry Contracting (OIC@unc.edu) to receive the dataset and codebook and agree to acknowledge NIH and the study investigators in any publications resulting from the data.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Label With Text Health Warning | Label With Pictorial Health Warning | Label With Neutral Statements About Vaping
Started | 456 | 457 | 456
Completed | 454 | 452 | 452
Not Completed | 2 | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Label With Text Health Warning | Label With Pictorial Health Warning | Label With Neutral Statements About Vaping | Total
Number analyzed (Participants) | 456 | 457 | 456 | 1369
Age, Customized [Count of Participants; unit: Participants]
  21-29 years | 133 | 130 | 141 | 404
  30-39 years | 170 | 159 | 166 | 495
  40-49 years | 100 | 100 | 95 | 295
  50+ years | 53 | 68 | 54 | 175
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 193 | 197 | 208 | 598
  Male | 249 | 237 | 221 | 707
  Nonbinary/Another gender | 14 | 23 | 27 | 64
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaskan Native | 5 | 4 | 3 | 12
  Asian | 54 | 25 | 39 | 118
  Black or African American | 78 | 77 | 74 | 229
  Hispanic | 32 | 51 | 46 | 129
  Middle Eastern or North African | 2 | 8 | 2 | 12
  Native Hawaiian or other Pacific Islander | 1 | 4 | 3 | 8
  White | 194 | 196 | 183 | 573
  Multiracial or another race or ethnicity | 90 | 91 | 106 | 287
  Missing | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 456 | 457 | 456 | 1369

OUTCOME MEASURES:

1. Primary Outcome: Mean Vaping Quit Intentions Score
Description: The primary outcome is vaping quit intentions measured by 3 survey items at 5 time points: post-labeling (Visit 1) and at 1, 2, 3, and 4 weeks (Visits 2-5). Study investigators will average the items to create a score for each time point and take an average across the time points. The range for this measure will be 1 to 5, with higher values indicating higher quit intentions.
Time Frame: Up to 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Label With Text Health Warning | Label With Pictorial Health Warning | Label With Neutral Statements About Vaping
Number analyzed (Participants) | 456 | 457 | 456
score on a scale | 2.5 (1.3) | 2.5 (1.1) | 2.2 (1.0)
Statistical Analysis 1: Comparison: Label With Text Health Warning vs Label With Neutral Statements About Vaping; Test type: Superiority; p < .001, General linear model
Statistical Analysis 2: Comparison: Label With Text Health Warning vs Label With Pictorial Health Warning; Test type: Superiority; p = .78, General linear model

2. Secondary Outcome: Mean Knowledge Score
Description: Knowledge of health harms from vaping will be measured by 5 survey items at 5 time points: post-labeling (Visit 1) and at 1, 2, 3, and 4 weeks (Visits 2-5). Study investigators will score each item for accuracy (correct or incorrect) and average the scores (% correct) for each time point and take an average across the time points. The range for this measure will be 0% to 100%, with higher values indicating more accurate knowledge).
Time Frame: Up to 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Label With Text Health Warning | Label With Pictorial Health Warning | Label With Neutral Statements About Vaping
Number analyzed (Participants) | 456 | 457 | 456
score on a scale | 0.6 (0.3) | 0.6 (0.3) | 0.4 (0.3)
Statistical Analysis 1: Comparison: Label With Text Health Warning vs Label With Neutral Statements About Vaping; Test type: Superiority; p < .001, General linear model
Statistical Analysis 2: Comparison: Label With Text Health Warning vs Label With Pictorial Health Warning; Test type: Superiority; p = .66, General linear model

3. Secondary Outcome: Mean Cognitive Elaboration Score
Description: Cognitive elaboration (thinking about the label) will be measured by 3 survey items at 4 time points: 1, 2, 3, and 4 weeks (Visits 2-5). Study investigators will average the items to create a score for each time point and take an average across the time points. The range for this measure will be 1 to 5, with higher values indicating more cognitive elaboration.
Time Frame: Up to 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Label With Text Health Warning | Label With Pictorial Health Warning | Label With Neutral Statements About Vaping
Number analyzed (Participants) | 395 | 385 | 383
score on a scale | 2.7 (0.9) | 2.9 (0.9) | 2.0 (0.8)
Statistical Analysis 1: Comparison: Label With Text Health Warning vs Label With Neutral Statements About Vaping; Test type: Superiority; p < .001, General linear model
Statistical Analysis 2: Comparison: Label With Text Health Warning vs Label With Pictorial Health Warning; Test type: Superiority; p < .001, General linear model

4. Secondary Outcome: Mean Perceived Likelihood of Illness Score
Description: Perceived likelihood of illness from vaping will be measured by 3 survey items at 5 time points: post-labeling (Visit 1) and at 1, 2, 3, and 4 weeks (Visit 2-5). Study investigators will average the items to create a score for each time point and take an average across the time points. The range for this measure will be 1 to 5, with higher values indicating higher perceived likelihood.
Time Frame: Up to 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Label With Text Health Warning | Label With Pictorial Health Warning | Label With Neutral Statements About Vaping
Number analyzed (Participants) | 456 | 457 | 456
score on a scale | 3.1 (0.8) | 3.1 (0.8) | 2.9 (0.9)
Statistical Analysis 1: Comparison: Label With Text Health Warning vs Label With Neutral Statements About Vaping; Test type: Superiority; p = .001, General linear model
Statistical Analysis 2: Comparison: Label With Text Health Warning vs Label With Pictorial Health Warning; Test type: Superiority; p = .95, General linear model

5. Secondary Outcome: Mean Negative Affect Score
Description: Negative affective reactions to the labels will be measured by 5 survey items at 5 time points: post-labeling (Visit 1) and at 1, 2, 3, and 4 weeks (Visits 2-5). Study investigators will average the items to create a score for each time point and take an average across the time points. The range for this measure will be 1 to 5, with higher values indicating more negative affect.
Time Frame: Up to 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Label With Text Health Warning | Label With Pictorial Health Warning | Label With Neutral Statements About Vaping
Number analyzed (Participants) | 456 | 457 | 456
score on a scale | 2.1 (0.9) | 2.3 (1.0) | 1.4 (0.6)
Statistical Analysis 1: Comparison: Label With Text Health Warning vs Label With Neutral Statements About Vaping; Test type: Superiority; p < .001, General linear model
Statistical Analysis 2: Comparison: Label With Text Health Warning vs Label With Pictorial Health Warning; Test type: Superiority; p < .001, General linear model

6. Secondary Outcome: Mean Attention Score
Description: Attention to the labels will be measured by 3 survey items at 4 time points: 1, 2, 3, and 4 weeks (Visits 2-5). Study investigators will average the items to create a score for each time point and take an average across the time points. The range for this measure will be 1 to 5, with higher values indicating greater attention.
Time Frame: Up to 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Label With Text Health Warning | Label With Pictorial Health Warning | Label With Neutral Statements About Vaping
Number analyzed (Participants) | 395 | 385 | 383
score on a scale | 3.1 (0.9) | 3.3 (0.9) | 2.8 (0.9)
Statistical Analysis 1: Comparison: Label With Text Health Warning vs Label With Neutral Statements About Vaping; Test type: Superiority; p < .0001, General linear model
Statistical Analysis 2: Comparison: Label With Text Health Warning vs Label With Pictorial Health Warning; Test type: Superiority; p < .001, General linear model

7. Secondary Outcome: Mean Information Seeking Score
Description: Information seeking about the harms of vaping will be measured by 1 survey item at 4 time points: 1, 2, 3, and 4 weeks (Visits 2-5). Study investigators will score responses (0 times=0, 1-2 times=1.5, 3-5 times=4, 6+ times=6) and take an average across the time points. The range for this measure will be 0 times to 6 times), with higher values indicating more information seeking.
Time Frame: Up to 4 weeks
Measure: Mean (Standard Deviation); unit: number of times sought information
Arm/Group | Label With Text Health Warning | Label With Pictorial Health Warning | Label With Neutral Statements About Vaping
Number analyzed (Participants) | 395 | 385 | 383
number of times sought information | 1.3 (1.3) | 1.4 (1.3) | 0.8 (1.0)
Statistical Analysis 1: Comparison: Label With Text Health Warning vs Label With Neutral Statements About Vaping; Test type: Superiority; p < .001, General linear model
Statistical Analysis 2: Comparison: Label With Text Health Warning vs Label With Pictorial Health Warning; Test type: Superiority; p = .4, General linear model

8. Secondary Outcome: Mean Number of Conversations in Past Week
Description: Number of conversations with others about the labels, health harms caused by vaping, and quitting vaping will be measured by 3 survey items at 4 time points: 1, 2, 3, and 4 weeks (Visits 2-5). Study investigators will average the items to create a score for each time point and take an average across the time points. The range for this measure will be 0 times to 100 times, with higher values indicating more conversations.
Time Frame: Up to 4 weeks
Measure: Mean (Standard Deviation); unit: number of conversations
Arm/Group | Label With Text Health Warning | Label With Pictorial Health Warning | Label With Neutral Statements About Vaping
Number analyzed (Participants) | 395 | 385 | 383
number of conversations | 1.5 (2.2) | 1.7 (2.1) | 1.2 (1.8)
Statistical Analysis 1: Comparison: Label With Text Health Warning vs Label With Neutral Statements About Vaping; Test type: Superiority; p = .03, General linear model
Statistical Analysis 2: Comparison: Label With Text Health Warning vs Label With Pictorial Health Warning; Test type: Superiority; p = .4, General linear model

9. Secondary Outcome: Mean Vaping Reinforcement Attitudes Score
Description: Positive vaping reinforcement attitudes will be measured by 3 survey items at 5 time points: post-labeling (Visit 1) and at 1, 2, 3, and 4 weeks (Visits 2-5). We will take an average across the time points. The range for this measure will be 1 to 5, with higher values indicating more positive vaping reinforcement attitudes.
Time Frame: Up to 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Label With Text Health Warning | Label With Pictorial Health Warning | Label With Neutral Statements About Vaping
Number analyzed (Participants) | 456 | 457 | 456
units on a scale | 4.1 (0.8) | 4.1 (0.8) | 4.2 (0.8)
Statistical Analysis 1: Comparison: Label With Text Health Warning vs Label With Neutral Statements About Vaping; Test type: Superiority; p = .61, General linear model
Statistical Analysis 2: Comparison: Label With Text Health Warning vs Label With Pictorial Health Warning; Test type: Superiority; p = .68, General linear model

10. Secondary Outcome: Mean Uncontrolled Vaping Score
Description: Subjective uncontrolled vaping (vaping more than the user prefers) will be measured by 3 survey items at 4 time points: 1, 2, 3, and 4 weeks (Visit 2-5). Study investigators will average the items to create a score for each time point and take an average across the time points. The range for this measure will be 1 to 5, with higher values indicating vaping that is more uncontrolled.
Time Frame: Up to 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Label With Text Health Warning | Label With Pictorial Health Warning | Label With Neutral Statements About Vaping
Number analyzed (Participants) | 395 | 385 | 383
score on a scale | 2.4 (0.9) | 2.4 (1.0) | 2.3 (1.0)
Statistical Analysis 1: Comparison: Label With Text Health Warning vs Label With Neutral Statements About Vaping; Test type: Superiority; p = .4, General linear model
Statistical Analysis 2: Comparison: Label With Text Health Warning vs Label With Pictorial Health Warning; Test type: Superiority; p = .5, General linear model

11. Secondary Outcome: Mean Number of Times Forgoing a Vape in Past Week
Description: Number of times forgoing a vape in the last week will be measured by 4 survey items at 4 time points: 1, 2, 3, and 4 weeks (Visits 2-5). Study investigators will score responses (never=0, 1 time=1, 2 times=2, 3-5 times=4, 6+ times=6), average the items to create a score for each time point, and take an average across the time points. The range for this measure will be 0 times to 6 times, with higher values indicating more forgoing.
Time Frame: Up to 4 weeks
Measure: Mean (Standard Deviation); unit: number of times forgoing a vape
Arm/Group | Label With Text Health Warning | Label With Pictorial Health Warning | Label With Neutral Statements About Vaping
Number analyzed (Participants) | 395 | 385 | 383
number of times forgoing a vape | 1.7 (1.6) | 1.7 (1.5) | 1.3 (1.4)
Statistical Analysis 1: Comparison: Label With Text Health Warning vs Label With Neutral Statements About Vaping; Test type: Superiority; p = .001, General linear model
Statistical Analysis 2: Comparison: Label With Text Health Warning vs Label With Pictorial Health Warning; Test type: Superiority; p = .9, General linear model

12. Secondary Outcome: Percent of Participants Who Made a Vaping Quit Attempt in Past 4 Weeks
Description: Made vaping quit attempt will be measured by 1 survey item (not vaping for 1 day or longer in the last week because they were trying to stop vaping) at 4 time points: 1, 2, 3, and 4 weeks (Visits 2-5). There will be an additional item (not vaping for 1 day or longer since the start of the study) at 4 weeks (Visit 5). Study investigators will score the items for any quit attempts: 0 (no quit attempts) or 1 (one or more quit attempt across the 4 weeks).
Time Frame: Up to 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Label With Text Health Warning | Label With Pictorial Health Warning | Label With Neutral Statements About Vaping
Number analyzed (Participants) | 456 | 457 | 456
Participants | 217 | 204 | 211
Statistical Analysis 1: Comparison: Label With Text Health Warning vs Label With Neutral Statements About Vaping; Test type: Superiority; Odds Ratio (OR) = .9, 95% CI 2-sided [.73 to 1.2]
Statistical Analysis 2: Comparison: Label With Text Health Warning vs Label With Pictorial Health Warning; Test type: Superiority; Odds Ratio (OR) = .9, 95% CI 2-sided [.69 to 1.2]

13. Secondary Outcome: Percent of Participants Who Successfully Quit Vaping
Description: Successful quitting of vaping during the trial will be measured by 1 survey item at 1 time point (participants' last survey, usually Visit 5). Study investigators will score the item for successful quitting: 0 (vaping on one or more of the last 7 days) or 1 (no vaping).
Time Frame: At 4 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Label With Text Health Warning | Label With Pictorial Health Warning | Label With Neutral Statements About Vaping
Number analyzed (Participants) | 456 | 457 | 456
percentage of participants | 7.2 | 7.4 | 3.7
Statistical Analysis 1: Comparison: Label With Text Health Warning vs Label With Neutral Statements About Vaping; Test type: Superiority; Odds Ratio (OR) = .5, 95% CI 2-sided [.3 to .9]
Statistical Analysis 2: Comparison: Label With Text Health Warning vs Label With Pictorial Health Warning; Test type: Superiority; Odds Ratio (OR) = 1, 95% CI 2-sided [.6 to 1.7]

14. Secondary Outcome: Mean Inaccurate Risk Perception Score
Description: Inaccurate risk perception of vaping (believing vaping is the same or more harmful than smoking cigarettes) will be measured by 1 survey item at 5 time points: post-labeling (Visit 1) and 1, 2, 3, and 4 weeks (Visits 2-5). Study investigators will score the item for accuracy (vaping less harmful than smoking cigarettes=correct; other answers=incorrect) and take an average across the time points. The range for this measure will be 0% (no correct answers) to 100% (all correct answers), with higher values indicating more accurate risk perceptions.
Time Frame: Up to 4 weeks
Measure: Mean (Standard Deviation); unit: proportion of correct answers
Arm/Group | Label With Text Health Warning | Label With Pictorial Health Warning | Label With Neutral Statements About Vaping
Number analyzed (Participants) | 456 | 457 | 456
proportion of correct answers | 0.42 (0.42) | 0.44 (0.43) | 0.48 (0.43)
Statistical Analysis 1: Comparison: Label With Text Health Warning vs Label With Neutral Statements About Vaping; Test type: Superiority; p = .02, General linear model
Statistical Analysis 2: Comparison: Label With Text Health Warning vs Label With Pictorial Health Warning; Test type: Superiority; p = .5, General linear model

15. Secondary Outcome: Mean Stigma Score
Description: Stigma (expecting the labels will cause social disapproval of vaping) will be measured by 3 survey items at 5 time points: post-labeling (Visit 1) and at 1, 2, 3, and 4 weeks (Visits 2-5). Study investigators will average the items to create a score for each time point and take an average across the time points. The range for this measure will be 1 to 5, with higher values indicating more stigma.
Time Frame: Up to 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Label With Text Health Warning | Label With Pictorial Health Warning | Label With Neutral Statements About Vaping
Number analyzed (Participants) | 456 | 457 | 456
score on a scale | 1.9 (0.8) | 2.0 (0.9) | 1.6 (0.7)
Statistical Analysis 1: Comparison: Label With Text Health Warning vs Label With Neutral Statements About Vaping; Test type: Superiority; p < .001, General linear model
Statistical Analysis 2: Comparison: Label With Text Health Warning vs Label With Pictorial Health Warning; Test type: Superiority; p = .004, General linear model

16. Secondary Outcome: Mean Smoking Quit Intentions Score
Description: Smoking quit intentions will be measured by 3 survey items at 5 time points: post-labeling (Visit 1) and 1, 2, 3, and 4 weeks (Visits 2-5). Study investigators will average the items to create a score for each time point and take an average across the time points. The construct will be assessed only among cigarette smokers. The range for this measure will be 1 to 5, with higher values indicating higher intentions.
Time Frame: Up to 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Label With Text Health Warning | Label With Pictorial Health Warning | Label With Neutral Statements About Vaping
Number analyzed (Participants) | 456 | 457 | 456
score on a scale | 2.4 (0.9) | 2.5 (0.9) | 2.3 (0.9)
Statistical Analysis 1: Comparison: Label With Text Health Warning vs Label With Neutral Statements About Vaping; Test type: Superiority; p = 0.3, General linear model
Statistical Analysis 2: Comparison: Label With Text Health Warning vs Label With Pictorial Health Warning; Test type: Superiority; p = 0.5, General linear model

17. Secondary Outcome: Percent of Participants Who Made a Smoking Quit Attempt in Past 4 Weeks
Description: Made smoking quit attempt will be measured by 1 survey item (not smoking for 1 day or longer in the last week because they were trying to stop smoking) at 4 time points: 1, 2, 3, and 4 weeks (Visits 2-5). There will be an additional item (not smoking for 1 day or longer since the start of the study) at 4 weeks (Visit 5). Study investigators will score the items for any quit attempts: 0 (no quit attempts) or 1 (at least one quit attempt across the 4 weeks).
Time Frame: Up to 4 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Label With Text Health Warning | Label With Pictorial Health Warning | Label With Neutral Statements About Vaping
Number analyzed (Participants) | 456 | 457 | 456
percentage of participants | 54.3 | 67.9 | 63.1
Statistical Analysis 1: Comparison: Label With Text Health Warning vs Label With Neutral Statements About Vaping; Test type: Superiority; Odds Ratio (OR) = 1.4, 95% CI 2-sided [.99 to 2.1]
Statistical Analysis 2: Comparison: Label With Text Health Warning vs Label With Pictorial Health Warning; Test type: Superiority; Odds Ratio (OR) = 1.8, 95% CI 2-sided [1.2 to 2.6]

ADVERSE EVENTS:
Time Frame: From the time of signing informed consent, through study completion, a total of up to 4 weeks.
Arm/Group | Label With Text Health Warning | Label With Pictorial Health Warning | Label With Neutral Statements About Vaping
All-Cause Mortality (participants affected / at risk) | 0/456 | 0/457 | 0/456
Serious Adverse Events (participants affected / at risk) | 0/456 | 0/457 | 0/456
Other Adverse Events (participants affected / at risk) | 0/456 | 0/457 | 0/456

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2025-07-08): https://cdn.clinicaltrials.gov/large-docs/82/NCT05714982/Prot_004.pdf
  • Statistical Analysis Plan (2024-06-24): https://cdn.clinicaltrials.gov/large-docs/82/NCT05714982/SAP_001.pdf
  • Informed Consent Form (2023-08-11): https://cdn.clinicaltrials.gov/large-docs/82/NCT05714982/ICF_003.pdf